CLINICAL TRIAL: NCT01786291
Title: Effects of Positive Airway Pressure Therapy on Exercise Parameters in Obstructive Sleep Apnea
Brief Title: PAP Therapy Sleep Apnea and Exercise
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, meral uyar, Associate Professor, University of Gaziantep
Other Study IDs: uyku-cpet-1
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; continuous positive airway pressure; cardiopulmonary exercise test; VE/VCO2
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CPAP compliant: CPAP (continuous positive airway pressure) compliant patients
- CPAP non-compliant: patients who did not use CPAP therapy

SUMMARY:
Positive airway pressure (PAP) therapy is generally offered to patients with obstructive sleep apnea. The investigators suggest that beneficial effects of PAP therapy is by preventing apneas and therefore reducing cardiac and pulmonary morbidities. The investigators sought to verify this by assessing cardiac and pulmonary function during exercise.

ELIGIBILITY:
Inclusion Criteria:

* obstructive sleep apnea diagnosed by polysomnography
* CPAP therapy indicated

Exclusion Criteria:

* obstructive or restrictive lung disease
* cardiac failure
* acute coronary syndrome
* inability to cycle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients newly diasgnosed with obstructive sleep apnea in whom CPAP therapy was indicated
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
peak oxygen uptake | 30-60 days

SECONDARY OUTCOMES:
ventilatory equivalent for carbon dioxide at anaerobic threshold | 30-60 days

CONTACTS AND LOCATIONS:
Overall Officials: Meral Uyar, Assoc Prof, Principal Investigator — University of Gaziantep; Nazan Bayram, Assis Prof, Principal Investigator — University of Gaziantep
Locations (1):
- University of Gaziantep, Faculty of Medicine, Dept. of Pulmonary Diseases, Gaziantep, Turkey (Türkiye)